CLINICAL TRIAL: NCT03399344
Title: Clinical Impact of Dedicated MR Staging of Ovarian Cancer
Acronym: MRStagingOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M17MRO
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will undergo an additional MRI, including a diffusion-weighted sequence, for assessing the extent of peritoneal carcinomatosis. Whether or not cytoreductive surgery is feasible will be scored using the peritoneal cancer index on diffusion-weighted magnetic resonance imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DW-MRI (Other): Patients with undergo an additional diffusion-weighted MRI in addition to the standard diagnostic work-up
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — In addition to the standard diagnostic work-up patients will receive an additional MRI scan 0-21 days prior to their scheduled surgery.

SUMMARY:
The only chance of cure for patients with advanced stage ovarian cancer is complete cytoreductive surgery (CRS). The only way to determine whether complete CRS can be achieved is by a laparoscopy. However, diffusion-weighted magnetic resonance imaging (DW-MRI) has a very high sensitivity to detect small volume malignant disease, making it a potentially suitable staging tool. Aim of this study is to determine the performance of DW-MRI for predicting whether complete CRS can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced stage (FIGO stage III or IV) ovarian cancer scheduled for primary or interval cytoreductive surgery
* Age >18 years
* Written and signed informed consent
* WHO 0-2
* Able to read and write Dutch

Exclusion Criteria:

* Patients with contraindications for MRI
* Patients with contraindications for CRS
* Known additional malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females with ovarian cancer
Enrollment: 270 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of DW-MRI to predict a complete cytoreductive surgery | 1 month
  Patients will undergo an additional MRI, besides their regular diagnostic workup, for assessing the extent of peritoneal carcinomatosis. Whether or not complete cytoreductive surgery is feasible will be determined on DW-MRI independently by two radiologists. The outcome wil be defined as the number of cytoreductive procedures correctly predicted by DW-DWI.

CONTACTS AND LOCATIONS:
Locations (1):
- NKI-AVL, Amsterdam, Netherlands